CLINICAL TRIAL: NCT01035658
Title: A Phase I/II Study of the Combination of Pazopanib and Liposomal Doxorubicin (Doxil) in Patients With Advanced Relapsed Platinum-Sensitive or Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Adenocarcinoma
Brief Title: Pazopanib/Doxil in Adv Relapsed Plat Sensitive or Resistant Ovarian, Fallopian or Primary Peritoneal Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on analyses in Phase I, the study did not advance to Phase II.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GYN 26
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Carcinoma
Keywords: Pazopanib; Doxil; Liposomal doxorubicin; Advanced relapsed; platinum-sensitive; platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pazopanib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Level 1 (Experimental): Systemic therapy with pazopanib and liposomal doxorubicin (Doxil). Single-agent pazopanib will be given for a 7 day run-in period, followed by a combination of pazopanib (400mg) and liposomal doxorubicin (40mg) administered in 28-day treatment cycles. Cycles will continue until disease progression, unacceptable toxicity or withdrawal.
  Interventions: Drug: Pazopanib; Drug: Doxil
- Dose Level -1 (Experimental): Systemic therapy with pazopanib and liposomal doxorubicin (Doxil). Single-agent pazopanib will be given for a 7 day run-in period, followed by a combination of pazopanib (400mg) and liposomal doxorubicin (30mg) administered in 28-day treatment cycles. Cycles will continue until disease progression, unacceptable toxicity or withdrawal.
  Interventions: Drug: Pazopanib; Drug: Doxil
- Dose Level 1 Sequential (Experimental): Systemic therapy with pazopanib and liposomal doxorubicin (Doxil). In this schedule, liposomal doxorubicin (30mg) was given on day 1, and pazopanib (400mg) was given days 3 - 26 of each 28 day cycle. Cycles will continue until disease progression, unacceptable toxicity or withdrawal.
  Interventions: Drug: Pazopanib; Drug: Doxil
- Dose Level 2 Sequential (Experimental): Systemic therapy with pazopanib and liposomal doxorubicin (Doxil). In this schedule, liposomal doxorubicin (40mg) was given on day 1, and pazopanib (400mg) was given days 3 - 26 of each 28 day cycle. Cycles will continue until disease progression, unacceptable toxicity or withdrawal.
  Interventions: Drug: Pazopanib; Drug: Doxil

INTERVENTIONS:
Drug: Pazopanib — All patients will begin treatment with a 7-day run in period of single-agent pazopanib. Patients will receive pazopanib orally days 1-28 of a 28 day cycle.
  Other Names: Systemic therapy
Drug: Doxil — Liposomal doxorubicin (Doxil) will be administered IV on day 1 of a 28-day treatment cycle
  Other Names: Systemic therapy; Liposomal doxorubicin

SUMMARY:
In this study, patients with relapsed or refractory ovarian cancer will receive treatment with pazopanib and liposomal doxorubicin (Doxil) until disease progression or unacceptable toxicity occurs. The Phase I portion will define the dose limiting toxicity (DLT) of pazopanib and liposomal doxorubicin when administered in combination. Once the maximum tolerated dose has been identified in the Phase I portion, the Phase II portion will evaluate efficacy and safety of this combination in the same patient population.

DETAILED DESCRIPTION:
In this study, patients with relapsed or refractory ovarian cancer will receive treatment with pazopanib and liposomal doxorubicin (Doxil) until disease progression or unacceptable toxicity occurs. The Phase I portion will define the dose limiting toxicity (DLT) of pazopanib and liposomal doxorubicin when administered in combination. Once the maximum tolerated dose has been identified in the Phase I portion, the Phase II portion will evaluate efficacy and safety of this combination in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of epithelial ovarian carcinoma (FIGO Stage II to IV), primary peritoneal cancer or fallopian tube.
2. One or 2 previous chemotherapy regimens for advanced ovarian cancer. At least one of these regimens must have contained a platinum agent.
3. Patients who are platinum-resistant (relapse <6 months after completing a platinum-containing regimen) or platinum sensitive (relapse ≥ 6 months after platinum-containing regimen) are eligible.
4. Radiographically documented progression per RECIST criteria (version 1.1) or progression of CA-125 during or subsequent to the last chemotherapy regimen.
5. Measurable disease (RECIST criteria) or evaluable disease with elevated CA-125 level. Patients with normal CT scans and elevated CA-125 levels as the only indication of disease are not eligible. ECOG performance status of 0 or 1.
6. Normal left ventricular ejection fraction (LVEF) according to institutional standards.
7. Adequate recovery from recent surgery. At least 1 week must have elapsed from the time of a minor surgery (with the exception of portacath placement); at least 4 weeks must have elapsed from the time of a major surgery.
8. Laboratory values as follows:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥9g/dL. Patients may not have received RBC transfusions within 7 days of screening assessment.
   * Platelets ≥100,000/L
   * AST or ALT must be <2.5 x ULN (concomitant elevations in bilirubin and AST/ALT >1.0 x ULN are not permitted).
   * Total bilirubin <1.5 x the institutional ULN (if Gilberts syndrome, direct bilirubin ≤1.5 x ULN)
   * International normalized ratio (INR) 1.2 and activated partial thromboplastin time (aPTT) 1.2 the ULN (except for patients receiving anti-coagulation therapy)
   * Cr ≤ 1.5 x ULN. If Cr >1.5 x ULN, then calculated creatinine clearance must be ≥50 mL/min
   * Urine protein creatinine (UPC) ratio ≤1.0 at screening OR Urine dipstick for proteinuria <2+ (patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate <1g of protein in 24 hours to be eligible).
9. Patients must be 18 years of age.
10. Life expectancy of ≥12 weeks.
11. Patient must be accessible for treatment and follow-up.
12. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.
13. Females of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), include a female who has had: a hysterectomy, a bilateral oophorectomy, a bilateral tubal ligation, or is post-menopausal. Patients not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be ≥45 years old, or in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value <40pg/mL. Patients using HRT must have experienced total cessation of menses for ≥1 year and be ≥45 years old, or have had documented evidence of menopause based on FSH and estradiol prior to the initiation of HRT.
14. Women of childbearing potential must have a negative serum or urine pregnancy test performed ≤14 days prior to start of treatment. Women of childbearing potential must use effective birth control measures during treatment. Acceptable contraceptive methods include: 1) an intrauterine device with a documented failure rate of ≤1% per year, 2) a vasectomized partner who is sterile prior to the patient"s entry and is the sole sexual partner for that female, 3) abstinence 14 days prior to study entry, throughout the dosing period, and for at least 21 days after the last dose of protocol therapy, 4) double-barrier contraception, or 5) oral contraception. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.

Exclusion Criteria:

1. Patients may not have received either investigational or marketed agents, which act by primary anti-angiogenic mechanisms (i.e. bevacizumab).
2. Prior treatment with liposomal doxorubicin.
3. Patients with brain metastases. (Baseline imaging required only if clinically indicated).
4. Patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
5. Patients with hemoptysis within 6 weeks of first dose of study drug.
6. Patients who are pregnant or breast feeding.
7. Impaired cardiac function including any of the following conditions within the past 6 months:

   * NYHA Class II, III or IV heart failure.
   * QTc prolongation or other significant ECG abnormalities.
   * Myocardial infarction or unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * History of sustained ventricular tachycardia.
8. Patients must not have taken any potent CYP3A4 inhibitors <= 14 days prior to enrollment including but not limited to:

   • ketoconazole, itraconazole, troleandomycin, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, amprenavir, nefazodone, fluvoxamine, diltiazem, verapamil, mibefradil, cimetidine, cyclosporine, and grapefruit juice.
9. Uncontrolled hypertension (systolic blood pressure [BP] >180 or diastolic BP >100mm Hg) or uncontrolled cardiac arrhythmias (Patients with hypertension controlled by antihypertensive therapies are eligible.)
10. History of cerebrovascular accident (CVA), MI within 12 months or venous thrombosis within 12 weeks. (Patients with previous history of venous thrombosis on a stable dose of anticoagulation are allowed.)
11. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
12. Inability to swallow whole tablets.
13. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g., active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection).
14. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
15. Use of any non-approved or investigational agent <= 30 days prior to administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
16. Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS >= 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T.Michael Numnum, MD, Study Chair — SCRI Development Innovations, LLC
Locations (4):
- United States (4):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Insitute, Orlando, Florida
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
Started | 5 | 8 | 3 | 6
Completed | 5 | 8 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential | Total
Number analyzed (Participants) | 5 | 8 | 3 | 6 | 22
Age, Continuous [Median (Full Range); unit: years] | 62 [51 to 69] | 74 [31 to 90] | 64 [51 to 64] | 57 [49 to 79] | 64 [31 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 3 | 6 | 22
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 3 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Pazopanib and Liposomal Doxorubicin
Description: The MTD of the drug combination will be determined as the highest dose at which ≤1 of 6 subjects experiences a Grade 3 or Grade 4 DLT according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
Time Frame: 18 months
Measure: Number; unit: mg
Groups:
- Phase 1: All patients in Phase I (this section contains the Maximum Tolerated Dose)
Arm/Group | Phase 1
Number analyzed (Participants) | 22
mg
  Pazopanib | 400
  Liposomal doxorubicin | 30

2. Primary Outcome: Phase I - Dose Limiting Toxicities
Description: As requested, this outcome measure reports the number of patients experiencing dose limiting toxicities (DLTs) in the Phase I portion of the study
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
Number analyzed (Participants) | 5 | 8 | 3 | 6
participants | 3 | 1 | 0 | 0

3. Primary Outcome: Phase II: Progression Free Survival
Description: Defined as from date of randomization until objective tumor progression or death. Response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) and CA-125 response in patients using the Rustin Criteria.
Time Frame: 18 months
Population: Per protocol, study did not proceed to phase II based on analyses from phase I. Therefore, Phase II outcomes (all outcomes other than determination of the MTD) were not evaluated and will not be posted.
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Phase II - Overall Survival of Patients With Relapsed/Refractory Ovarian Cancer Following Treatment With Pazopanib and Liposomal Doxorubicin
Time Frame: 18 months
Population: as for outcome 3
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Response Rate in the Subsets of Patients With Platinum-sensitive and Platinum-refractory Ovarian Carcinoma
Description: The response rate in the subsets of patients with platinum-sensitive and platinum-refractory ovarian carcinoma is evaluated as a measure of efficacy of pazopanib/liposomal doxorubicin. Response rate ( Percentage of patients whose disease decreased (Partial response - PR) and/or disappears (Complete response - CR) after treatment) was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) and CA-125 response in patients using the Rustin Criteria. CR: disappearance of all target and nontarget lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Normalization of CA125, if elevated at baseline, is required for ovarian carcinoma studies. PR is >= 30% decrease in the sum of longest diameter(LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of nontarget lesions and no new lesions.
Time Frame: 18 months
Population: Two patients stopped treatment prior to first reevaluation and hence were not included in the analysis. one patient's Recurrence status is unknown and thus was not evaluable
Measure: Count of Participants; unit: Participants
Groups:
- Platinum Refractory Disease; Platinum Sensitive Disease: Systemic therapy with pazopanib and liposomal doxorubicin (Doxil). Single-agent pazopanib will be given for a 7 day run-in period, followed by a combination of pazopanib (400mg) and liposomal doxorubicin (40mg) administered in 28-day treatment cycles. Cycles will continue until disease progression, unacceptable toxicity or withdrawal.
Arm/Group | Platinum Refractory Disease | Platinum Sensitive Disease
Number analyzed (Participants) | 8 | 11
Participants | 3 | 5

6. Secondary Outcome: Number of Participants Experiencing Adverse Events With the Combination of Pazopanib and Liposomal Doxorubicin Doses
Description: An adverse event (AE) is the development of an undesirable medical condition, or the deterioration of a pre-existing medical condition (other than the condition that is being treated by the trial) following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. The number of participants experiencing such adverse events that are possibly/probably/definitely related to the study drugs are reported here.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
Number analyzed (Participants) | 5 | 8 | 3 | 6
Participants | 5 | 7 | 2 | 6

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1 Sequential | Dose Level 2 Sequential
All-Cause Mortality (participants affected / at risk) | 4/5 | 7/8 | 3/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/8 | 2/3 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level -1 (N=8) | Dose Level 1 Sequential (N=3) | Dose Level 2 Sequential (N=6)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, disease progression (General disorders) | 0 | 1 | 0 | 0
Infections and infestations - Other, pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level -1 (N=8) | Dose Level 1 Sequential (N=3) | Dose Level 2 Sequential (N=6)
White blood cell decreased (Investigations) | 2 | 5 | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 3 | 1 | 3
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 3
Platelet count decreased (Investigations) | 0 | 3 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 1
Fatigue (General disorders) | 3 | 4 | 3 | 3
Nausea (Gastrointestinal disorders) | 4 | 3 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 1 | 2
Mucositis (Gastrointestinal disorders) | 3 | 2 | 0 | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
General disorders and administration site conditions - Other, hemorrhage (General disorders) | 0 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
Per protocol, study did not proceed to phase II based on analyses from phase I. Therefore, Phase II outcomes (all outcomes other than determination of the MTD) were not evaluated and will not be posted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites